CLINICAL TRIAL: NCT04244045
Title: Effect of Adding Sub-occipital Muscle Inhibition Technique Versus Slump Stretch Position to Passive Hamstring Stretch on Hamstring Flexibility in Patients With Short Hamstring Syndrome
Brief Title: Sub Occipital Muscle Inhibition Versus Slump Stretch Position in Short Hamstring Syndrome Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jouf University (Other)
Collaborators: Cairo University (Other); Olfat Ibrahim Ali (Unknown); Alaa Mohamed Al abbas (Unknown); Sara Hamed Elzarea (Unknown)
Responsible Party: Principal Investigator, Hadaya Mosaad, lecturer, Jouf University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/002566
Record Dates: First submitted 2020-01-22; First posted 2020-01-28 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Musculoskeletal Diseases or Conditions
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental group 1 (Experimental): suboccipital muscle inhibition plus passive stretch of hamstring muscle.
  Interventions: Other: Suboccipital muscle inhibition
- Experimental group 2 (Experimental): Neural slump strtch position plus passive stretch of hamstring muscle.
  Interventions: Other: Suboccipital muscle inhibition
- Control group (Active Comparator): passive stretch of hamstring muscle
  Interventions: Other: Suboccipital muscle inhibition

INTERVENTIONS:
Other: Suboccipital muscle inhibition — The patient was asked to flex his hip joint with complete knee extension and ankle in neutral position. The therapist stretches the hamstring of the dominant side; distal hand of the therapist on planter surface of foot for dorsiflexion. and proximal hand on the knee to increase the length of the muscle, maintain this stretching for 60 seconds then relax .Sub occipital muscle inhibition:
  The Patient is supine, The therapist stretch the sub occipital, flexes the head of the patient to get the chin to the manibiurim sternii, maintaining this position for 60seconds then relax Slump strtch position:Patient in comfortable short sitting position at the edge of the bed with the trunk in an millitary straight position then ask the patient to slump the flex his neck and street the knee joint in complete extension the at the end of the procedure do active dorsiflexion at the tested foot
  Other Names: slump stretch position; Passive stretch of the hamstring muscle.

SUMMARY:
45 female participants with short hamstring syndrome were devided into one of the three groups; Group I: suboccipital muscle inhinbition plus passive hamstring stretch, group II: Slump stretch position plus Passive hamstring stretch, and group III: Passive stretch of hamstring muscle. Assessment methods were Straight leg raising test, forward flexion test and popliteal angle test, were measured at baseline, immediately after 1st treatment session then after 4 weeks of treatment.

DETAILED DESCRIPTION:
Forty five university undergraduate female students volunteered to participate in the study, age = 18-25 years old, body mass index 18-25 kg/cm square.

All subjects were free from injury or disease expected to affect hamstring length or ability to perform the exercises Design of the study was single-blind randomized clinical trial. The subjects were randomly assigned in to one of the three methods of treatment, which are group 1 (study group1): suboccipital muscle inhibition plus passive stretch of hamstring muscle, Group II: ( Study groupII): received neural slump test position plus passive stretch of hamstring muscle, Group III (control group): received only passive stretch of hamstring muscle.

Treatment Procedures:

Passive stretching of hamstring muscle:

Patient in comfortable supine lying position and therapist stride standing beside the dominant side of the patient. The patient was asked to flex his hip joint with complete knee extension and ankle in neutral position. The therapist stretches the hamstring of the dominant side; distal hand of the therapist on planter surface of foot for dorsiflexion to increase flexibility of hamstring muscle and proximal hand on the knee to increase the length of the muscle, maintain this stretching for 60 seconds then relax (8)

Sub occipital muscle inhibition:

The Patient is in comfortable supine lying position with eye closed - for more relaxation- and the head out of the bed resting on therapist hand to manipulate the sub occipital area. The therapist stretch the sub occipital, flexes the head of the patient to get the chin to the manibiurim sternii, maintaining this position for 60seconds then relax (9)

Neural dynamic slump stretch:

Patient in comfortable short sitting position at the edge of the bed with the trunk in an millitary straight position then ask the patient to slump the flex his neck and street the knee joint in complete extension the at the end of the procedure do active dorsiflexion at the tested foot .(10)

ELIGIBILITY:
Inclusion Criteria:

1. Being females.
2. Age between 18-28 years old.
3. BMI: 18-25 kg/square meter.
4. All subjects were free from injury or disease expected to affect hamstring length or ability to perform the exercises.
5. Straight leg raising test (SLR) is less than 80 degree from supine position.
6. Popliteal angle test, operationally defined by a knee flexion angle greater than 15˚ as measured by a screening exam using active knee extension in supine with hip flexed 90˚

Exclusion Criteria:

* Hamstring injury within the past year.
* Exceeding 80° in the initial SLR test. Popleteal knee angle less than 15 degree. -
* Verbal report of performing regular lower extremity. Muscle stretching exercises.
* History of neck trauma (whiplash). Neck symptoms.-
* History of recent fracture in any part of the body.
* History of growth disorders,

Ages: 18 Years to 28 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Straight leg raising test | after 4 weeks of intervention.
  the patient was supine lying position with hip and knee extension at the starting position, then the patient was asked to actively flex hip joint as much as possible while maintaining the knee in extension position. Then with the goniometer the therapist started to determine the angle of hip flexion, patients were excluded if the SRL was more than 80˚at the initial evaluation

SECONDARY OUTCOMES:
Popliteal Angle Test | after 4 weeks of intervention.
  while the patient was in supine line position, the hip and knee joint was flexed to 90˚ then the patient was asked to extend the knee joint as much as possible with maintaining the hip in flexion 90˚. Then with the goniometer the therapist determines the angle of the knee flexion, subjects were excluded if their angle of flexion less than 15 ˚
Forward flexion test | after 4 weeks of treatment.
  the patient was stride standing on footstep facing the therapist and then asked to flex her trunk with his hands facing forward, maintaining the knee in extended position. The therapist then measures the distance between the middle finger and the ground while the trunk is in complete flexion.

CONTACTS AND LOCATIONS:
Overall Officials: Hadaya M El Adl, Phd, Study Director — Jouf University, Collage of applied medical science.
Locations (1):
- Faculty of physical therapy, Cairo University., Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Informed consent form, Study protocol
Supporting Information: Study Protocol, SAP, ICF
Time Frame: we will share results after 6 months of publication.